CLINICAL TRIAL: NCT02144350
Title: Hyperbaric Oxygen Therapy for Moderate to Severe Ulcerative Colitis Flares: A Multi-center Randomized Double Blind Sham Controlled Trial
Brief Title: Hyperbaric Oxygen for Ulcerative Colitis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Mayo Clinic (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Corey Siegel, Section Chief, Section of Gastroenterology, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Broad-IBD-0372
Record Dates: First submitted 2014-05-13; First posted 2014-05-22 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2016-11

CONDITIONS: Ulcerative Colitis
Keywords: hyperbaric oxygen
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): patients will undergo daily hyperbaric oxygen sessions in addition to IV steroids for 10 days.
  Interventions: Procedure: Hyperbaric oxygen
- Sham (Sham Comparator): Patients will undergo sham hyperbaric air sessions in addition to IV steroids for 10 days
  Interventions: Procedure: Sham Hyperbaric Air

INTERVENTIONS:
Procedure: Hyperbaric oxygen — patients will be placed in a monoplane chamber and pressurized to 2.4 atmospheres with 100% oxygen for 90 minutes per session.
  Arms: Intervention
Procedure: Sham Hyperbaric Air — Patients will undergo a brief compression to 1.34 atmospheres with room air and then they will be brought back to 1.1 atmospheres to complete a 90 minute session.
  Arms: Sham

SUMMARY:
The investigators aim to prospectively study the feasibility and clinical impact of hyperbaric oxygen therapy in acute hospitalized moderate to severe ulcerative colitis flares as an adjunct to standard medical treatment. Specifically, we will investigate the impact of hyperbaric oxygen therapy on clinical response/remission and serum and mucosal inflammatory markers. The investigators expect that hyperbaric oxygen therapy will improve patient responsiveness to steroids and avoid progression to second line therapy during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* known or newly diagnosed moderate to severe ulcerative colitis with a Mayo score of greater than 6
* Mayo endoscopic sub-score of greater than or equal to 2
* Risk score of greater than or equal to 4 points

Exclusion Criteria:

* Complication requiring urgent surgical intervention (in the opinion of the investigators)

Clinically significant cardiac, renal, neurological, endocrine, respiratory or hepatic impairment in the opinion of the investigator, including but not limited to:

* Pulmonary i. COPD with CO2 retention; Previous/current imaging showing hyperinflation/air trapping/bullous disease/blebs (opinion of investigators) ii. Current pneumothorax or previous spontaneous pneumothorax iii. Bronchogenic cyst(s)
* Cardiac i. Uncontrolled HTN (systolic >160 or diastolic >100) ii. Unstable angina or myocardial infarction within the previous 3 months iii. Ejection fraction < 35% iv. Current or previous amiodarone use v. ICD in place vi. Pacemaker in place not approved for chamber use
* Hematological/Oncological i. Current chemotherapeutic drug use, and past history of bleomycin use. ii. Hereditary Spherocytosis iii. Sickle cell anemia
* Gastrointestinal and Infectious Disease i. Known or suspected Crohn's disease ii. Previous infection with mycobacterium, fungus, HIV, Hepatitis B or C iii. Gastrointestinal or systemic infection including, but not limited to, --Clostridium difficile iv. Current capsule endoscopy or previously non-retrieved capsule Endocrinology i. Uncontrolled hyperthyroidism

Neurological and Psychological i. Vagal or other nerve stimulators

ii. Uncontrolled seizure disorder

iii. Medications or medical conditions that lower seizure threshold (in the opinion of the investigator) iv. Drug or alcohol abuse/dependence v. Current treatment for alcohol cessation with disulfiram vi. Current or recent (within past week) use of baclofen Head and Neck i. Previous middle ear damage, surgery or infection(s) which may increase the risk for needing ear tubes (in the opinion of the investigator) ii. Current or previous retinal detachment or optic neuritis iii. Retinal or vitreous surgery within the past 3 months Miscellaneous i. Implanted devices not on the approved list for use with HBOT

Women who are pregnant or nursing. Women with childbearing potential were required to use effective birth control if not surgically sterile or postmenopausal for >2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Primary Response | Day 5
  Impact of hyperbaric oxygen therapy on clinical response/remission to medical therapy as measured by the partial Mayo score at study day 5. Clinical remission will be defined as a partial Mayo score of less than or equal to 2 with no individual sub-score exceeding 1 point. Clinical response will be defined as a decrease in partial Mayo score greater than or equal to 2 points with a decrease in rectal bleeding sub-score of greater than or equal to 1 point, or an absolute rectal bleeding sub-score of 0 or 1.

SECONDARY OUTCOMES:
Reduction in Full Mayo Score | Day 10
  We will compare the % and absolute reduction in the full Mayo score at study day 10 between the intervention and sham control group
Reduction in Inflammatory Markers | Day 10
  We will compare the % and absolute reduction in the CRP and ESR at study days 3, 5 and 10 between the intervention and sham control group
Progression to Second Line Therapy | Day 10
  We will compare the proportion of patients requiring infliximab, cyclosporine or colectomy during hospitalization between the intervention and sham control group

OTHER OUTCOMES:
Hyperbaric Oxygen Safety | before and after hyperbaric oxygen treatments
  The rate of barotrauma, seizures, or claustrophobia with hyperbaric oxygen therapy will be monitored to ensure there are no safety concerns with this intervention. Patients will be assessed before and after each treatment session for any complications related to hyperbaric oxygen therapy. This will be done daily until all 10 treatments are completed.

CONTACTS AND LOCATIONS:
Overall Officials: Corey A Siegel, MD, MS, Study Director — Dartmouth-Hitchcock Medical Center
Locations (3):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Pittsburgh, Pittsburgh, Pennsylvania